CLINICAL TRIAL: NCT04494399
Title: An Open-label Randomised Controlled Trial on IFN Beta-1b and Ribavirin Combination, as Treatment for Covid-19 Infection
Brief Title: IFN Beta-1b and Ribavirin for Covid-19
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UW 20-513
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Covid19
Keywords: interferon beta-1b; ribavirin; hospitalised; patients
MeSH Terms: conditions — COVID-19 | interventions — Interferon beta-1b; Ribavirin

STUDY DESIGN:
Intervention Model Description: open label randomised controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): 5-day course of daily subcutaneous injection of interferon β-1b 2mL (16 million IU) consecutively and oral ribavirin 400mg twice daily plus standard care
  Interventions: Drug: Interferon beta-1b; Drug: Ribavirin
- Control group (No Intervention): Standard care alone

INTERVENTIONS:
Drug: Interferon beta-1b — 5-day course of daily subcutaneous injection of interferon β-1b 16 million IU
  Arms: Treatment group
Drug: Ribavirin — 5-day course of oral ribavirin 400mg twice daily
  Arms: Treatment group

SUMMARY:
As of 1 July 2020, more than 10 million people been confirmed to have infected by SARS-CoV-2, resulting in more than 500,000 deaths. No specific antiviral treatment for the SARS-CoV-2 is currently available, but existing medication could be repurposed.

The investigators therefore propose to conduct an open-label randomized controlled trial on a short course of interferon β-1b and ribavirin combination treatment for patients hospitalized for COVID-19 infection.

DETAILED DESCRIPTION:
The novel coronavirus (SARS-CoV-2), is a single-stranded RNA coronavirus. The virus was first isolated from patients presented with pneumonia in Wuhan in December 2019. It is believed that the virus first emerged from patients working in the Wuhan Seafood Market which also sold contaminated wild animals, consumed as a local delicacy. Sequences of the Wuhan betacoronavirus show similarities to betacoronaviruses found in bats, sharing a common ancestor with the 2003 SARS coronavirus (SARS-CoV).

The SARS-CoV-2 has since spread from China to the rest of the world. As of 1 July 2020, more than 10 million people been confirmed to have infected by SARS-CoV-2, resulting in more than 500,000 deaths. No specific antiviral treatment for the SARS-CoV-2 is currently available, but existing medication could be repurposed.

Previously, the investigators have demonstrated that interferon beta-1b, commonly used in the treatment of multiple sclerosis and lopinavir/ ritonavir, also demonstrated to improve the outcome of MERS-CoV infection in a non-human primate model of common marmoset. More recently, the investigators have demonstrated that the triple combination of interferon β-1b, lopinavir/ ritonavir and ribavirin was significantly more effective in alleviating symptoms and respiratory SARS-CoV-2 viral load than lopinavir/ ritonavir with ribavirin or lopinavir/ ritonavir alone, suggesting that interferon β-1b might be the most potent antiviral among the three and lopinavir/ ritonavir is associated with relatively more side effects including diarrhoea and cardiac arrhythmia.

Therefore, the investigators propose to conduct an open-label randomized controlled trial on a short course of interferon β-1b and ribavirin combination treatment for patients hospitalized for COVID-19 infection.

Patients will be randomly assigned to one of the two groups: the Treatment group: a 5-day course of subcutaneous injection of interferon β-1b 2mL (16 million IU) consecutively and oral ribavirin 400mg twice daily, or the Control group: supportive care alone (1:1).

For patients randomized to the Control group, if the nasopharyngeal swab (NPS) or throat saliva (TS) viral load is still detectable on day 3, the patients will receive the same treatment as in the Treatment group from day 4 to day 8.

ELIGIBILITY:
Inclusion Criteria:

1. Recruited subjects include all adult patients ≥18 years hospitalized for virologic confirmed SARS-CoV-2 infection.
2. All subjects give written informed consent. For patients who are critically ill, requiring ICU, ventilation or confused, informed consent will be obtained from spouse, next-of-kin or legal guardians.
3. Subjects must be available to complete the study and comply with study procedures. Willingness to allow for serum samples to be stored beyond the study period, for potential additional future testing to better characterize immune response.

Exclusion Criteria:

1. Inability to comprehend and to follow all required study procedures.
2. Allergy or severe reactions to the study drugs
3. Patients taking medication that will potentially interact with l interferon beta-1b or ribavirin
4. Pregnant or lactation women
5. Patients with known history of severe depression
6. Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to recruitment in this study or expect to receive an experimental agent during this study.
7. To participate in an unrelated trial during the current clinical trial. Nevertheless, the patients have the right to withdraw from the current clinical trial to join another clinical trial.
8. Have a history of alcohol or drug abuse in the last 5 years.
9. Have any condition that the investigator believes may interfere with successful completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical symptoms alleviation | 7 days
  Time to complete alleviation of symptoms as defined by NEWS2 of 0 maintained for 24 hours

SECONDARY OUTCOMES:
Hospitalisation | 14 days
  Length of hospitalisation
Time to negative viral load | 7 days
  Time to negative nasopharyngeal swab and throat saliva viral load by RT-PCR
Inflammatory changes | 7 days
  Cytokine/ chemokine changes
Mortality | 30 days
  One month mortality rate
Adverse events and serious adverse events | 30 days
  Adverse events and serious adverse events within 30 days of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ivan FN Hung, MD FRCP, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Background] Hung IF, Lung KC, Tso EY, Liu R, Chung TW, Chu MY, Ng YY, Lo J, Chan J, Tam AR, Shum HP, Chan V, Wu AK, Sin KM, Leung WS, Law WL, Lung DC, Sin S, Yeung P, Yip CC, Zhang RR, Fung AY, Yan EY, Leung KH, Ip JD, Chu AW, Chan WM, Ng AC, Lee R, Fung K, Yeung A, Wu TC, Chan JW, Yan WW, Chan WM, Chan JF, Lie AK, Tsang OT, Cheng VC, Que TL, Lau CS, Chan KH, To KK, Yuen KY. Triple combination of interferon beta-1b, lopinavir-ritonavir, and ribavirin in the treatment of patients admitted to hospital with COVID-19: an open-label, randomised, phase 2 trial. Lancet. 2020 May 30;395(10238):1695-1704. doi: 10.1016/S0140-6736(20)31042-4. Epub 2020 May 10. PMID 32401715
- [Background] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Background] Chu H, Chan JF, Wang Y, Yuen TT, Chai Y, Hou Y, Shuai H, Yang D, Hu B, Huang X, Zhang X, Cai JP, Zhou J, Yuan S, Kok KH, To KK, Chan IH, Zhang AJ, Sit KY, Au WK, Yuen KY. Comparative Replication and Immune Activation Profiles of SARS-CoV-2 and SARS-CoV in Human Lungs: An Ex Vivo Study With Implications for the Pathogenesis of COVID-19. Clin Infect Dis. 2020 Sep 12;71(6):1400-1409. doi: 10.1093/cid/ciaa410. PMID 32270184
- [Background] Chan JF, Yao Y, Yeung ML, Deng W, Bao L, Jia L, Li F, Xiao C, Gao H, Yu P, Cai JP, Chu H, Zhou J, Chen H, Qin C, Yuen KY. Treatment With Lopinavir/Ritonavir or Interferon-beta1b Improves Outcome of MERS-CoV Infection in a Nonhuman Primate Model of Common Marmoset. J Infect Dis. 2015 Dec 15;212(12):1904-13. doi: 10.1093/infdis/jiv392. Epub 2015 Jul 21. PMID 26198719
- [Background] Yuan S, Chan CC, Chik KK, Tsang JO, Liang R, Cao J, Tang K, Cai JP, Ye ZW, Yin F, To KK, Chu H, Jin DY, Hung IF, Yuen KY, Chan JF. Broad-Spectrum Host-Based Antivirals Targeting the Interferon and Lipogenesis Pathways as Potential Treatment Options for the Pandemic Coronavirus Disease 2019 (COVID-19). Viruses. 2020 Jun 10;12(6):628. doi: 10.3390/v12060628. PMID 32532085
- [Background] Blanco-Melo D, Nilsson-Payant BE, Liu WC, Uhl S, Hoagland D, Moller R, Jordan TX, Oishi K, Panis M, Sachs D, Wang TT, Schwartz RE, Lim JK, Albrecht RA, tenOever BR. Imbalanced Host Response to SARS-CoV-2 Drives Development of COVID-19. Cell. 2020 May 28;181(5):1036-1045.e9. doi: 10.1016/j.cell.2020.04.026. Epub 2020 May 15. PMID 32416070